CLINICAL TRIAL: NCT06424964
Title: Use of Long-Acting Injectable Cabotegravir/Rilpivirine for the Treatment of HIV in Belgium
Status: Recruiting | Type: Observational
Sponsor: Belgian Research on AIDS and HIV Consortium (Other)
Responsible Party: Principal Investigator, Rakan Nasreddine, Head of Research, Belgian Research on AIDS and HIV Consortium
Other Study IDs: 2024/1-12
Record Dates: First submitted 2024-05-14; First posted 2024-05-22 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This will be a multi-center, single arm observational cohort study with an assessment of patient-reported outcomes (PROs) and of clinical and virologic outcomes.

Primary outcome • Evaluate patient perception of, and satisfaction with, long-acting injectable (LAI) cabotegravir/rilpivirine (CAB/RPV) for the treatment of HIV

Secondary outcomes

• Description of the demographic, HIV-, and non-HIV-related characteristics of participants included in this analysis

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 patients, aged 18 years and above, having received at least 1 dose of LAI CAB/RPV between September 1, 2021, and March 31, 2024.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited at one of the participating HIV reference centers (HRCs). These centers are part of the 12 official HIV treatment centers in Belgium and work in concert as members of the Belgian Research on AIDS & HIV Consortium (BREACH).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate participant perception of, and satisfaction with, LAI CAB/RPV for the treatment of HIV | Within the first 12 weeks of the study
  Participants will be asked to complete a 32-item paper questionnaire relating to their HIV treatment of LAI CAB/RPV. Questions will focus on how their daily life and quality of life has been affected by switching to LAI CAB/RPV. The questionnaire that will be used is not a standardized questionnaire but rather a questionnaire that was developped by the study team.

SECONDARY OUTCOMES:
Proportion of participants with virologic suppression at months 5 and 11 after initiation of LAI CAB/RPV | Months 5 and 11
Proportion of participants that experience loss of virologic suppression by month 11 | Month 11
Description of HIV resistance-associated mutations that are present at the time of loss of virologic suppression | Month 11
  If a participant experiences loss of virologic suppression, then if an HIV resistance test was performed at that time, the resistance-associated mutations observed will be reported.
Proportion of participants with a viral blip at months 5 and 11 | Months 5 and 11
Change, from baseline, of CD4+ T-cell count and CD4+/CD8+ ratio at months 5 and 11 | Months 5 and 11
Proportion of participants that are adherent to treatment at months 5 and 11 | Months 5 and 11
  LAI CAB/RPV must be taken every two months, which therefore requires that a target date be specified in advance of when the next treatment injection should be. This measure will evaluate the proportion of participants that presented to their clinic to receive their treatment either on the target date or within 7 days after (this will be considered adherent) and the proportion of participants that received their treatment more than 7 days after their target date (this will be considered non adherent)
Proportion of participants that discontinue their treatment over the study period | Month 11
Incidence of discontinuation of treatment over the study period | Month 11
  This measure will be reported in person/years
Reasons for discontinuation of treatment over the study period | Month 11
  This measure will report all the reasons for which participants discontinued their treatment
Time to discontinuation of treatment over the study period | Month 11
  This measure will be reported by median time to discontinuation (months) and inter-quartile range
Proportion of participants that experience injection-site reactions (ISRs) and acceptability of ISRs | Within the first 12 weeks of the study
Change in weight from baseline and a ≥10% weight gain from baseline at months 5 and 11 | Months 5 and 11
Proportion of participants that become hepatitis B virus (HBV) seropositive at months 5 and 11 | Months 5 and 11

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane De Wit, MD/PhD, Principal Investigator — Belgian Research on AIDS & HIV Consortium
Locations (1):
- Saint-Pierre University Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No